CLINICAL TRIAL: NCT05558982
Title: Phase II Trial of BXCL701 and Pembrolizumab in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: BXCL701 and Pembrolizumab in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: EXPEL PANC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: BioXcel Therapeutics Inc (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005453
Record Dates: First submitted 2022-09-02; First posted 2022-09-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — PT-100 dipeptide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BXCL701 plus Pembrolizumab (Experimental)
  Interventions: Drug: BXCL701; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BXCL701 — BXCL701 0.3 mg, orally, twice a day on days 1-14 every 21 days
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenous (IV) on day 1 every 21 days.
  Other Names: Keytruda

SUMMARY:
Single-arm, open label study to determine the 18 week progression-free survival rate of the combination of BXCL701 and pembrolizumab in patients with pancreatic ductal adenocarcinoma in the second-line metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed pancreatic ductal adenocarcinoma with metastatic disease (mixed histology is acceptable as long adenocarcinoma is the dominant histological subtype)
* Patient must consent to two mandatory biopsies and have tumor amenable to serial core biopsies
* Measurable disease by iRECIST v. 1.1 criteria (tumor ≥ 1 cm in longest diameter on axial image on CT or MRI and/or lymph node(s) ≥ 1.5 cm in short axis on CT or MRI) on baseline imaging
* Documented progression of disease or intolerance on at least one regimen for metastatic disease (progression during or within 3 months of the completion of adjuvant therapy is acceptable)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2 (see Table 2)
* Age ≥ 18 years
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery (SRS) at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intracranial disease
* Patients with available standard 12-lead ECG with the following parameters at screening (defined as the mean of the triplicate ECGs):

  o QTcB (Bazett's formula) interval at screening <480msec
* Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥100 × 109/L; hemoglobin ≥ 8.0 g/dL (with no prior red blood cell transfusions during the prior 14 days)
* Renal function: serum creatinine ≤ 1.5 × upper normal limit of institution's normal range or creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
* Hepatic function: AST and ALT ≤ 3.0 × the upper normal limit of institution's normal range. Total bilirubin ≤ 1.5 × the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT < 5 × the upper normal limit of institution's normal range, and total bilirubin >1.5 - 3.0 x the upper normal limit of institution's normal range are acceptable as long as there is no persistent nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia.
* Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring "Twilight" sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator.
* Women of childbearing potential must have a negative serum pregnancy test during the screening period and on C1D1 and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient is capable of swallowing pills whole.
* Patient is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
* Patient's acute toxic effects of previous anticancer therapy have resolved to ≤ Grade 1 except for Grade 2-3 peripheral neuropathy or any grade of alopecia.
* Male patients and their female partners of childbearing potential must agree and commit to use a barrier contraception (e.g., condom with spermicidal foam/gel/film/cream/ suppository) throughout the duration of the study until at least 6 months following the last dose of study drug, in addition to their female partners using either an intrauterine device or hormonal contraception and continuing until at least 6 months following the last dose of study drug. This criterion may be waived for male patients who have had a vasectomy >6 months before signing the informed consent form.

Exclusion Criteria:

* Patients previously exposed to FAP inhibitors, DPP inhibitors, or monoclonal antibodies targeting anti-PD-1, anti-PD-L1, or anti-CTLA-4.
* Prior anti-tumor therapy within 2 weeks of C1D1 (defined as, but not limited to, anti-cancer agents (cytotoxic chemotherapy, immunotherapy, and biologic therapy), radiotherapy, and investigational agents), the "washout period."
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic symptomatic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial, or viral infection).
* Women who are pregnant or breastfeeding.
* Psychiatric illness or social situation that would limit compliance with study requirements.
* Concurrent malignancy or malignancy within 2 years prior to C1D1, with the exception of adequately treated cutaneous basal or squamous cell carcinoma, non-melanomatous skin cancer, curatively resected cervical cancer, or any locally treated malignancy deemed low likelihood for recurrence or metastasis by the investigator.
* Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient has a known history of HIV infection or chronic, active hepatitis B or C (testing is not mandatory) - patients with hepatitis C status-post treatment with undetectable viral load are eligible.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Patient has uncontrolled, clinically significant pulmonary disease (e.g. chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the investigator would put the patient at significant risk for pulmonary complications during the study.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
  * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
  * Inability to determine the QT interval on screening
* Patients with history of symptomatic orthostatic hypotension within 3 months prior to enrollment, defined as a drop in systolic blood pressure (SBP) of ≥ 20 mmHg or diastolic blood pressure (DBP) of ≥ 10 mmHg with assumption of an upright posture.
* Patients with a history of (non-infectious) pneumonitis that required steroids, current pneumonitis, or those who have a history of interstitial lung disease.
* Patients who have received a live-virus vaccination within 30 days of planned treatment start date.
* Patient must not have active known or suspected autoimmune disease requiring systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (e.g., celiac disease) are permitted to enroll.
* Patient must not have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses ≤10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 18 weeks | 18 weeks

SECONDARY OUTCOMES:
Incidence of Adverse events | From start of intervention until 30 days following discontinuation of intervention
  Adverse events as per CTCAE v. 5.0
Objective response rate | Through study completion, on average 18 weeks
  Objective response by iRECIST v. 1.1
Median Duration of response (DOR) | 24 months
Median Progression-free survival (PFS) | 24 months
Median Overall survival (OS) | 24 months
Change in tumor marker (CA19-9) | Through study completion, on average 18 weeks
  Best change in tumor marker

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weinberg, MD, Study Chair — Georgetown University
Locations (3):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No